CLINICAL TRIAL: NCT02848599
Title: The Influence of Postoperative Analgesia on Systemic Inflammatory Response and Postoperative Cognitive Disfunction in Elderly Patients After Surgical Repair of Femoral Fractures
Brief Title: The Influence of Postoperative Analgesia on Systemic Inflammatory Response and POCD After Femoral Fractures Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-1:6563-3/2014
Record Dates: First submitted 2016-07-20; First posted 2016-07-28 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: postoperative analgesia; postoperative cognitive disfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Morphine; Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- morphine (Active Comparator): The patient-controlled intravenous analgesia with morphine (basal flow of 0.5-2 mg / h, bolus dose of 0.5 mg, lockout interval of 20 minutes, hour limit of 3 doses), which will be carried out 72 hours after the surgery
  Interventions: Drug: morphine
- levobupivacaine (Active Comparator): Upon completion of the operation for a period of 72 hours will be implemented continuous epidural local anesthetic through the Patient Controlled Analgesia (PCA) pump (Levobupivacaine 0.125%, basal flow of 6 ml / hour, a bolus dose of 2 ml, lockout interval of 20 minutes, hour limit of 3 doses).
  Interventions: Drug: levobupivacaine

INTERVENTIONS:
Drug: morphine
  Arms: morphine
Drug: levobupivacaine
  Other Names: Chirocaine
  Arms: levobupivacaine

SUMMARY:
The purpose of this study is to determine whether epidural levobupivacaine applied for the purpose of post-operative analgesia compared to systemic analgesia with morphine leads to better pain control, stronger suppression of the inflammatory response and the production of inflammatory mediators, faster recovery of patients and consequently less incidence of postoperative cognitive dysfunction (POCD) in elderly patients after surgical treatment of femoral fractures.

DETAILED DESCRIPTION:
The research will be carried out at the Department of Surgery at Clinical Hospital Centre(CHC) Osijek after approval by the Ethics Committee of CHC Osijek and will be organized as a prospective randomized trial. Respecting the including and excluding criteria for participation in the study, the research will include 70 patients aged 65 years and over who are undergoing surgery for proximal femur fractures and will be operated with the same operating technique (osteosynthesis with nail). All participants will receive the same type of anesthesia and one of two forms of post-operative analgesia, so it will be divided into two groups (35 patients) depending on which form of post-operative analgesia receive. Randomization will be performed by drawing an envelope in which the specified one or other form of post-operative analgesia will be written. The study will be stopped in case of serious complications life-threatening (excessive sedation, respiratory insufficiency, hemodynamic instability and profound hypotension, heart rhythm disorders), which could possibly be related to the administration of drugs used for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* patients age 65 and over
* fracture of the proximal femur
* preoperative assessment American Society of Anesthesiologists(ASA) score I - ASA III
* a written consent of the patient to participate in research

Exclusion Criteria:

* patient non-compliance
* ASA status IV and IV above
* patients younger than 65 years
* dementia, Parkinson's disease, cerebrovascular accident history; simultaneous head injuries,the use of opioids and benzodiazepines longer than a month before the surgery; alcoholism; serious liver disease (class C according to Child-Pugh's classification); severe kidney disease that require dialysis
* result of MMSE test (Mini-Mental State Examination) under 17
* the existence of any contraindications for the implementation of regional anesthesia and one or other form of post-operative analgesia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Kristek, MD, Principal Investigator — Clinical Hospital Centre Osijek
Locations (1):
- Clinical Hospital Centre Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Raats JW, van Eijsden WA, Crolla RM, Steyerberg EW, van der Laan L. Risk Factors and Outcomes for Postoperative Delirium after Major Surgery in Elderly Patients. PLoS One. 2015 Aug 20;10(8):e0136071. doi: 10.1371/journal.pone.0136071. eCollection 2015. PMID 26291459
- [Background] Wang W, Wang Y, Wu H, Lei L, Xu S, Shen X, Guo X, Shen R, Xia X, Liu Y, Wang F. Postoperative cognitive dysfunction: current developments in mechanism and prevention. Med Sci Monit. 2014 Oct 12;20:1908-12. doi: 10.12659/MSM.892485. PMID 25306127
- [Background] Vega P E, Nazar J C, Rattalino F M, Pedemonte T J, Carrasco G M. [Postoperative delirium among older people]. Rev Med Chil. 2014 Apr;142(4):481-93. doi: 10.4067/S0034-98872014000400010. Spanish. PMID 25117039
- [Background] Vacas S, Degos V, Feng X, Maze M. The neuroinflammatory response of postoperative cognitive decline. Br Med Bull. 2013;106(1):161-78. doi: 10.1093/bmb/ldt006. Epub 2013 Apr 4. PMID 23558082
- [Background] Zywiel MG, Prabhu A, Perruccio AV, Gandhi R. The influence of anesthesia and pain management on cognitive dysfunction after joint arthroplasty: a systematic review. Clin Orthop Relat Res. 2014 May;472(5):1453-66. doi: 10.1007/s11999-013-3363-2. PMID 24186470
- [Background] Kampe S, Weinreich G, Darr C, Eicker K, Stamatis G, Hachenberg T. The impact of epidural analgesia compared to systemic opioid-based analgesia with regard to length of hospital stay and recovery of bowel function: retrospective evaluation of 1555 patients undergoing thoracotomy. J Cardiothorac Surg. 2014 Nov 23;9:175. doi: 10.1186/s13019-014-0175-8. PMID 25417134
- [Background] Popping DM, Elia N, Van Aken HK, Marret E, Schug SA, Kranke P, Wenk M, Tramer MR. Impact of epidural analgesia on mortality and morbidity after surgery: systematic review and meta-analysis of randomized controlled trials. Ann Surg. 2014 Jun;259(6):1056-67. doi: 10.1097/SLA.0000000000000237. PMID 24096762
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Background] Hansen MV. Chronobiology, cognitive function and depressive symptoms in surgical patients. Dan Med J. 2014 Sep;61(9):B4914. PMID 25186550
- [Background] Seitz DP, Adunuri N, Gill SS, Rochon PA. Prevalence of dementia and cognitive impairment among older adults with hip fractures. J Am Med Dir Assoc. 2011 Oct;12(8):556-564. doi: 10.1016/j.jamda.2010.12.001. Epub 2011 Mar 8. PMID 21450227
- [Background] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557
- [Background] van Harten AE, Scheeren TW, Absalom AR. A review of postoperative cognitive dysfunction and neuroinflammation associated with cardiac surgery and anaesthesia. Anaesthesia. 2012 Mar;67(3):280-93. doi: 10.1111/j.1365-2044.2011.07008.x. PMID 22321085
- [Background] Cunningham C. Systemic inflammation and delirium: important co-factors in the progression of dementia. Biochem Soc Trans. 2011 Aug;39(4):945-53. doi: 10.1042/BST0390945. PMID 21787328
- [Background] Steinman L. Modulation of postoperative cognitive decline via blockade of inflammatory cytokines outside the brain. Proc Natl Acad Sci U S A. 2010 Nov 30;107(48):20595-6. doi: 10.1073/pnas.1015282107. Epub 2010 Nov 22. No abstract available. PMID 21098269
- [Background] Peng L, Xu L, Ouyang W. Role of peripheral inflammatory markers in postoperative cognitive dysfunction (POCD): a meta-analysis. PLoS One. 2013 Nov 13;8(11):e79624. doi: 10.1371/journal.pone.0079624. eCollection 2013. PMID 24236147
- [Background] Rade MC, Yadeau JT, Ford C, Reid MC. Postoperative delirium in elderly patients after elective hip or knee arthroplasty performed under regional anesthesia. HSS J. 2011 Jul;7(2):151-6. doi: 10.1007/s11420-011-9195-2. Epub 2011 Feb 11. PMID 22754416
- [Background] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Background] Wang Y, Sands LP, Vaurio L, Mullen EA, Leung JM. The effects of postoperative pain and its management on postoperative cognitive dysfunction. Am J Geriatr Psychiatry. 2007 Jan;15(1):50-9. doi: 10.1097/01.JGP.0000229792.31009.da. PMID 17194815
- [Background] Zura M, Kozmar A, Sakic K, Malenica B, Hrgovic Z. Effect of spinal and general anesthesia on serum concentration of pro-inflammatory and anti-inflammatory cytokines. Immunobiology. 2012 Jun;217(6):622-7. doi: 10.1016/j.imbio.2011.10.018. Epub 2011 Nov 3. PMID 22217966
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Derived] Kristek G, Rados I, Kristek D, Kapural L, Neskovic N, Skiljic S, Horvat V, Mandic S, Harsanji-Drenjancevic I. Influence of postoperative analgesia on systemic inflammatory response and postoperative cognitive dysfunction after femoral fractures surgery: a randomized controlled trial. Reg Anesth Pain Med. 2019 Jan;44(1):59-68. doi: 10.1136/rapm-2018-000023. PMID 30640654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2016 to September 2017, 86 patients were included in the study in accordance with the inclusion criteria and 70 of them completed the study. The study design was a prospective, randomized, controlled trial. It was conducted at the University Hospital Osijek (Croatia).
Pre-assignment Details: No patients were excluded from the study before assignment to groups.
Groups:
- Morphine: The patient-controlled intravenous analgesia with morphine (basal flow of 0.5-2 mg / h, bolus dose of 0.5 mg, lockout interval of 20 minutes, hour limit of 3 doses), which will be carried out 72 hours after the surgery
  morphine
- Levobupivacaine: Upon completion of the operation for a period of 72 hours will be implemented continuous epidural local anesthetic through the Patient Controlled Analgesia (PCA) pump (Levobupivacaine 0.125%, basal flow of 6 ml / hour, a bolus dose of 2 ml, lockout interval of 20 minutes, hour limit of 3 doses).
  levobupivacaine
Period: Overall Study
Arm/Group | Morphine | Levobupivacaine
Started | 42 | 44
Completed | 35 | 35
Not Completed | 7 | 9
Not completed — Protocol Violation | 7 | 9

BASELINE CHARACTERISTICS:
Population: The reasons for exclusion of 16 patients were: inability to perform combined spinal-epidural anaesthesia (5 patients), technical problems with PCA pump (4 patients), withdrawal of epidural catheter (2 patients), postoperative delirium and use of antipsychotics (3 patients) and fever and use of antipyretics (2 patients).
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Levobupivacaine | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 35 | 35 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants]
  No school | 1 | 1 | 2
  Less than high school | 31 | 29 | 60
  High school | 3 | 5 | 8
ASA (American Society of Anesthesiologist physical status) [Count of Participants; unit: Participants] — ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA II | 3 | 3 | 6
    ASA III | 32 | 32 | 64
Duration of surgery [Median (Inter-Quartile Range); unit: minutes] | 49 [45 to 68] | 52 [44 to 66] | 52 [45 to 68]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 24.8 [21.5 to 29.8] | 23.9 [21.6 to 26.9] | 24.4 [21.6 to 27.8]
Perioperative transfusion [Median (Inter-Quartile Range); unit: Units of PRBC (packed red blood cells)] — Units of PRBC (packed red blood cells) given.
  Units of PRBC (packed red blood cells) | 2 [0 to 2] | 2 [0 to 2] | 2 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Interleukin-6 Concentration in Peripheral Blood.
Description: Measurement will be done before and 24 and 72 hours after the surgery.
Time Frame: Before, 24 and 72 hours after the surgery
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Morphine | Levobupivacaine
Number analyzed (Participants) | 35 | 35
pg/ml
  Before surgery | 27.2 [17.8 to 46.8] | 26.6 [19.7 to 38]
  24h after surgery | 104 [73 to 156.8] | 97.7 [65.9 to 119.1]
  72h after surgery | 50 [30.2 to 97.5] | 30.5 [23.1 to 52.4]

2. Primary Outcome: Changes in Cognitive Function
Description: Assessment of cognitive function will be done using the Mini-mental state examination (MMSE) rating scales before and 24,48,72,96 and 120 hours after the surgery at the same time every morning.
  Mini-Mental State Examination Scale: minimum score is 0 and maximum score is 30; the severity of cognitive impairment: no cognitive impairment=25-30; mild cognitive impairment=19-24; moderate cognitive impairment=10-18; and severe cognitive impairment<9. Higher scores mean a better and lower scores mean a worse outcome.
Time Frame: Before, 24,48,72,96 and 120 hours after the surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Morphine: 35 participants who received morphine iv
- Levobupivacaine: 35 participants who received 0,125% levobupivacaine epiduraly
Arm/Group | Morphine | Levobupivacaine
Number analyzed (Participants) | 35 | 35
score on a scale
  Before surgery | 21 [19 to 23] | 22 [20 to 25]
  24 h after surgery | 20 [18 to 23] | 22 [20 to 25]
  48 h after surgery | 20 [18 to 23] | 21 [20 to 24]
  72 h after surgery | 20 [17 to 23] | 21 [20 to 25]
  96 h after surgery | 20 [15 to 23] | 21 [20 to 25]
  120 h after surgery | 20 [17 to 23] | 22 [20 to 25]

3. Secondary Outcome: Changes in C-reactive Protein (CRP) Levels
Description: Measurement will be done before and 24,72 and 120 hours after the surgery.
Time Frame: Before, 24,72 and 120 hours after the surgery
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Morphine | Levobupivacaine
Number analyzed (Participants) | 35 | 35
mg/L
  Before surgery | 57.2 [10 to 90.3] | 57.8 [36.7 to 70.2]
  24 h after surgery | 106.2 [74.1 to 145] | 98.1 [77.1 to 116.8]
  72 h after surgery | 118.5 [82.9 to 149.9] | 95 [71.2 to 117.9]
  120 h after surgery | 66.9 [40.6 to 98.2] | 54.6 [30.7 to 70]

4. Secondary Outcome: Changes in Fibrinogen Concentrations in Peripheral Blood
Description: Measurement will be done before and 24,72 and 120 hours after the surgery.
Time Frame: Before, 24,72 and 120 hours after the surgery
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Morphine | Levobupivacaine
Number analyzed (Participants) | 35 | 35
g/L
  Before surgery | 5.5 [4.8 to 6.1] | 4.5 [3.8 to 5.3]
  24 h after surgery | 5.3 [4.8 to 5.6] | 4.7 [3.9 to 5.2]
  72 h after surgery | 5.7 [5.4 to 6.4] | 5.2 [4.4 to 6.2]
  120 h after surgery | 5.4 [4.7 to 6] | 5 [4.2 to 5.4]

5. Secondary Outcome: Changes in Pain Intensity
Description: Assessment will be done using Numeric Rating Scale (NRS). During the first 72 hours after the surgery assessment will be done every 3 hours, after that assessment will be done 3 times daily. Median of 8 time points measurements during the first 24, 48 and 72 hours after the surgery will be reported. After that, median of 3 time points will be reported from the 4. to 6. postoperative day and on the day of discharge.
  Minimum score 0 and maximum score 10 ( 0-No Pain; 1-3 Mild Pain; 4-6 Moderate Pain; 7-10 Severe Pain ). Higher scores mean a worse and lower scores mean a better outcome.
Time Frame: During the first 72 hours after the surgery assessment will be done every 3 hours, after that assessment will be done 3 times daily until discharge
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Morphine | Levobupivacaine
Number analyzed (Participants) | 35 | 35
score on a scale
  3,6,9,12,15,18,21 and 24h after surgery | 1.4 [0.6 to 2.9] | 0.6 [0.3 to 0.9]
  27,30,33,36,39,42,45 and 48h after surgery | 1.5 [0.8 to 2.3] | 0.5 [0.3 to 0.9]
  51,54,57,60,63,66,69 and 72h after surgery | 1.4 [0.9 to 1.9] | 0.5 [0.1 to 0.8]
  4. postoperative day (every 8 hours) | 1.4 [0.8 to 1.9] | 0.3 [0 to 0.8]
  5. postoperative day (every 8 hours) | 1.4 [1 to 2] | 0 [0 to 1]
  6. postoperative day (every 8 hours) | 1.3 [0.7 to 2.3] | 0 [0 to 0.7]
  Day of discharge | 1 [0 to 1] | 0 [0 to 0]

6. Secondary Outcome: Postoperative Hospital Stay
Description: Duration of postoperative hospital stay in days
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Morphine | Levobupivacaine
Number analyzed (Participants) | 42 | 44
days | 7 [7 to 8] | 7 [7 to 8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from end of the surgery until discharge from the hospital or date of death from any cause, whichever came first, assessed up to 10 days.
Description: Gastrointestinal side effects- nausea, constipation, vomiting Neurological side effects- paresthesia
Arm/Group | Morphine | Levobupivacaine
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 5/35 | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=35) | Levobupivacaine (N=35)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02848599/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02848599/SAP_001.pdf